CLINICAL TRIAL: NCT03404908
Title: Postoperative Analgesia With Transversus Abdominis Plane Block or Quadratus Lumborum Block in Patients After Cesarian Delivery
Brief Title: TAP vs QLB in Patients After Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/238/2017
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cesarean Section; Postoperative Pain
Keywords: transversus abdominis plane block; quadratus lumborum block; neuropathic pain
MeSH Terms: conditions — Pain, Postoperative; Neuralgia | interventions — Ropivacaine; Needles; Acetaminophen; Dipyrone; Ketoprofen; Morphine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP (Experimental): Ultrasound-guided transversus abdominis plane block at the end of cesarean section
  Interventions: Procedure: TAP (transversus abdominis plane block); Drug: Ropivacaine; Device: Needle; Drug: paracetamol; Drug: metamizole; Drug: Ketoprofen; Drug: Morphine
- QLB (Experimental): Ultrasound-guided quadratus lumborum block at the end of cesarean section
  Interventions: Procedure: QL (quadratus lumborum block); Drug: Ropivacaine; Device: Needle; Drug: paracetamol; Drug: metamizole; Drug: Ketoprofen; Drug: Morphine

INTERVENTIONS:
Procedure: TAP (transversus abdominis plane block) — the ultrasound-guided regional block of abdominal wall muscles to treat acute postoperative pain. Stimuplex Ultra 360 needle will be used and 0.375% ropivacaine administered (0.2 mL/kg).
  Arms: TAP
Procedure: QL (quadratus lumborum block) — the ultrasound-guided regional block of abdominal wall muscles to treat acute pain, similar to transversus abdominis plane block, but with a distribution of local anesthetic towards paravertebral space. Stimuplex Ultra 360 needle will be used and 0.25% bupivacaine administered (0.2 mL/kg).
  Arms: QLB
Drug: Ropivacaine — In both groups (TAP&QLB) 0.375% ropivacaine will be given (0.2 mL/kg)
Device: Needle — Ultrasound-guided, Stimuplex ultra 360 needle will be used in the study
Drug: paracetamol — Intravenous paracetamol will be used (1.0 gram), up to 4 grams per day
Drug: metamizole — Intravenous metamizole will be used (1.0 gram), up to 4 grams per day
Drug: Ketoprofen — Intravenous ketoprofen will be used (0.1 gram), up to 200 milligrams per day
Drug: Morphine — Intravenous morphine (5 mg) will be given when pain exceeds 40 mm in VAS (maximum 2 doses per day)

SUMMARY:
Comparison of two types of analgesia after cesarean section All patients will be anesthetized with spinal technique. Ultrasound-guided transversus abdominis plane or quadratus lumborum block to treat postoperative pain. Postoperative pain will be measured with visual-analog scale (VAS). 1, 2, 6 months after surgery each patient will be called to assess neuropathic pain with Neuropathic Pain Symptom Inventory (NPSI).

DETAILED DESCRIPTION:
Written consent will be obtained before the cesarean section. Only subarachnoidally anesthetized patients may participate in the study. Pencil-point spinal needle and bupivacaine (Marcaine Heavy Spinal 0.5 %) will be used.

At the end of surgery ultrasound-guided regional block will be performed. Each patient will be randomly allocated to one of the treated group: transversus abdominis plane block (TAP) or quadratus lumborum (QL). Patients receive 0.2 mL of local anesthetic solution (0.375 % ropivacaine) on each side.

Postoperative pain will be measured with VAS (visual-analog scale) 2, 4, 8, 12 and 24 hours after the end of the operation.

Paracetamol, metamizole, ketoprofen may be given as required. Whenever pain exceeds 40 (VAS) 5 mg of morphine will be given intravenously (maximum two dosages per day).

1, 3, 6 months patients will be called to assess neuropathic pain. Neuropathic Pain Symptom Inventory (NPSI) will be used.

ELIGIBILITY:
Inclusion Criteria:

* obtained consent
* singleton pregnancy
* subarachnoid anesthesia

Exclusion Criteria:

* coagulopathy
* allergy to local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — parturients
Enrollment: 105 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | up to 24 hours after the surgery
  Acute pain measured with VAS (visual-analogue scale). VAS in milimmeters. Minimum value 0, maximum 100. Less better - less severe pain. 0 no pain at all.

SECONDARY OUTCOMES:
Neuropathic pain | 6 months from the surgery
  Neuropathic pain occurrence assessed with Neuropathic Pain Symptom Inventory (NPSI) 10 descriptive variables, each one from 0 to 10. 0 means no pain. 10 very high chance of occurrence of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mirosław Czuczwar, M.D., PhD, Study Chair — Medical University of Lublin
Locations (1):
- II Department of Anesthesia and Intensive Care, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No